CLINICAL TRIAL: NCT06146153
Title: Impact of Various Palatal Vault Configurations of Edentulous Arches on Scan Accuracy. An Invivo Clinical Study
Brief Title: Intra Oral Scanning of Edentulous Arches
Status: Completed | Type: Observational
Sponsor: October University for Modern Sciences and Arts (Other)
Responsible Party: Principal Investigator, Dina ElAwady, Associate professor, October University for Modern Sciences and Arts
Other Study IDs: MSA University
Record Dates: First submitted 2023-11-18; First posted 2023-11-24 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Edentulous Jaw
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Class I: (medium U-vault)
  Interventions: Diagnostic Test: digital impression
- Class II: (deep-vault)
  Interventions: Diagnostic Test: digital impression
- Class III: flat vault
  Interventions: Diagnostic Test: digital impression

INTERVENTIONS:
Diagnostic Test: digital impression — intra oral scanning

SUMMARY:
the aim of this study is to compare the influence of different palatal vault configurations on the accuracy and scan speed of IO scans in cases of completely edentulous arches. The null hypothesis is that there is no difference in scanning time, and trueness and precision of IO scans between class I, II and III palatal vault configurations.

DETAILED DESCRIPTION:
A reference model will be created for each of the three groups with different palatal vault configurations. PVS material (DMG Silagum, Germany) will be used for impressions in a one-step process by an experienced operator, and type IV plaster (Heraeus, Germany) will be used to produce the models. These models will then bedigitized by an experienced operator using an extraoral scanner (Trios 3; 3Shape, Copenhagen, Denmark). The STL scan file of the maxillary model will be imported into CAD software (Meshmixer; Autodesk, San Rafael, CA, USA) to generate a reference file. Reference markers will then be added to the digital files to aid the superimposition process during digital subtraction operations.For intraoral scans, the entire maxilla of each patient will be digitally captured using an intraoral scanner (TRIOS POD, 3Shape, Copenhagen, Denmark).According to ISO standards, specifically ISO 5725-1, the accuracy of digital impressions obtained with intraoral scanners (IOS) will be evaluated according to two main parameters: trueness and precision.

ELIGIBILITY:
Inclusion Criteria:

* 1. Full tooth loss in the maxilla; 2. Absence of infectious diseases; 3. Systemic good health; 4. Age between 50 and 75 years; 5. Willingness to cooperate throughout the data collection process

Exclusion Criteria:

* Exclusion criteria included: 1. Presence of any remaining teeth; 2. Inability to comprehend the study's objectives and procedures; 3. Palatal defect or lesion; 4. Postoperative scarring on the palate; 5. Limitations in mouth opening.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All eligible participants who will comprehend the study's purpose and expresse their willingness to take part and sign a consent form will be enrolled in the study. The subjects will consist of dental patients who were seeking treatment for complete tooth loss in either the upper or lower jaw, or both. A total of thirty patients with complete edentulism, attending the outpatient clinic of MSA University, will be recruited for this research.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Trueness | 15 days
  Trueness is the degree of agreement between the digital impression and the reference scan. To assess trueness, we will measure the deviation between the reference and scanned files

SECONDARY OUTCOMES:
precision | 15 days
  Precision, is a statistical measure that quantifies the level of similarity between repeated samples within the same group. In the context of this study, the IOS impression STL files will be compared to each other in a manner similar to the previous comparisons

CONTACTS AND LOCATIONS:
Overall Officials: Dina Elawady, A.Prof, Principal Investigator — MSA University
Locations (1):
- MSA University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No